CLINICAL TRIAL: NCT00538720
Title: Pilot Study to Detect and Assess the Effect of Vitamin D Replacement on Gland Size by 4DCT in Patients With Primary Hyperparathyroidism (PHPT)
Brief Title: Effects of Vitamin D Replacement in Patients With Primary Hyperparathyroidism (PHPT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-0425; NCI-2012-01591 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; PHPT; Parathyroid glands; Vitamin D deficiency; Vitamin D; Ergocalciferol
MeSH Terms: conditions — Hyperparathyroidism; Hyperparathyroidism, Primary; Vitamin D Deficiency | interventions — Vitamin D; Ergocalciferols; Four-Dimensional Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Experimental): Vitamin D starting dose 50,000 IU by mouth 3 times weekly for three weeks (+/- one week), then 50,000 IU twice weekly for 6 weeks (+/- one week).
  Interventions: Drug: Vitamin D; Device: Four-dimensional computed tomography (4DCT)

INTERVENTIONS:
Drug: Vitamin D — Starting dose 50,000 IU by mouth 3 times weekly for three weeks (+/- one week), then 50,000 IU twice weekly for 6 weeks (+/- one week).
  Other Names: Ergocalciferol
Device: Four-dimensional computed tomography (4DCT) — Four-dimensional computed tomography (4DCT) scan of the neck.
  Other Names: 4DCT; 4-D Computed Tomography

SUMMARY:
The goal of this clinical research study is to learn how the standard practice of giving Vitamin D supplements to patients with a Vitamin D deficiency may affect the size of the parathyroid glands in patients with PHPT and a Vitamin D deficiency.

DETAILED DESCRIPTION:
The Study Vitamin:

In patients with PHPT and a Vitamin D deficiency, Vitamin D supplements are routinely given to bring Vitamin D blood levels up to a normal level before surgery on any abnormal parathyroid glands. When patients have Vitamin D deficiency, they do not absorb calcium very well, so the parathyroid glands have to work harder. This may cause the parathyroid glands to become larger.

Baseline:

If you are found to be eligible to take part in this study, as part of your routine standard of care, you will have a 4-dimensional computed tomography (4DCT) scan of the neck. This 4DCT will be used to find the size and location of your parathyroid glands to help the surgeon in planning the surgery.

Vitamin D Administration:

You will receive Vitamin D pills to take at home, by mouth. You should take the Vitamin D at the same time each day. If it causes an upset stomach, you should take it with food.

You will be given a study diary to record the days that you take the Vitamin D pills. You will return the diary at the end of each cycle.

Cycle 1:

During Cycle 1 (about the first 3 weeks of the study, +/- 1 week), you will take 3 Vitamin D pills per week about every other day (for example, Mondays, Wednesdays, and Fridays).

At the end of Cycle 1, blood (about 1 teaspoon) will be drawn to check Vitamin D levels.

If your Vitamin D level is not high enough at this first Cycle 1 study visit, you will repeat the Cycle 1 dosing schedule a second time. At the end of this second Cycle 1 dosing schedule, you will have another blood test (about 1 teaspoon) to check your Vitamin D levels. If your Vitamin D level is not high enough, you will be taken off study.

If your Vitamin D level is high enough after either your first or second Cycle 1 dosing schedule, you will go to Cycle 2.

Cycle 2:

During Cycle 2, the dosing schedule for Vitamin D is 2 pills per week for 6 weeks (+/- 1 week). You should try to take the pill on the same day of the week.

At the end of Cycle 2, blood (about 1 teaspoon) will be drawn to check Vitamin D levels.

If your Vitamin D level is not high enough at this first Cycle 2 study visit, you will repeat the Cycle 2 dosing schedule a second time. At the end of this second Cycle 2 dosing schedule, you will have another blood test (about 1 teaspoon) to check your Vitamin D levels. If your Vitamin D level is not high enough, you will be taken off study.

If your Vitamin D level is high enough after either your first or second Cycle 2 dosing schedule, you will go to Cycle 3.

Cycle 3:

During Cycle 3, the dosing schedule for Vitamin D is 2 pills per week for 6 weeks (+/- 1 week).

At the end of Cycle 3, blood (about 1 teaspoon) will be drawn to check Vitamin D levels.

If your Vitamin D level is high enough, you will have another 4DCT scan of your neck, for the purpose of this research study. This second scan will be used to see if your parathyroid glands have changed in size. Before this second scan, blood (about 1/2 teaspoon) will be drawn to check your kidney function.

If your Vitamin D level is not high enough, you will be taken off study.

Routine Surgical Treatment:

Within 3 weeks after your second 4DCT scan, your routine surgery for PHPT will be performed. You will sign a separate consent form and its risks will be described in more detail at that time. Your removed parathyroid glands will examined.

Length of Study:

Your active participation in this study will be over after you have surgery. If the side effects of PHPT indicate that you may need to have parathyroid surgery earlier, you will be taken off study early and have the surgery as soon as possible.

This is an investigational study. Vitamin D supplements are commercially available and FDA approved for use in patients with PHPT and a Vitamin D deficiency to bring the Vitamin D blood levels to normal before surgery. It is considered experimental to have a second 4DCT scan after your Vitamin D levels are high enough.

Up to 22 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with PHPT (inappropriate PTH level in the setting of a high or high-normal corrected serum calcium level equal to or greater than 10.0 mg/dL)
2. Be considered an appropriate surgical candidate
3. Be older than 21 years of age
4. Have a vitamin D (25-OHD) level less than or equal to 20ng/ml
5. Female participants of childbearing potential must have a negative pregnancy test (urinary or serum beta-HCG) within two weeks before signing consent

Exclusion Criteria:

1. Have any other functional tumors if they have familial multiple endocrine neoplasia syndrome 1 or 2 (MEN 1 or MEN 2)
2. Have a corrected calcium level greater than 13mg/dL
3. Have a recent history of kidney stones
4. Have a recent history of pancreatitis
5. Have a recent history of cardiac arrhythmia (eg atrial fibrillation)
6. Unable to keep still for 2 minutes without coughing
7. Having a body habitus that prevents adequate images to be obtained through the region of the parathyroids (ie typically weighing in excess of 250Lbs)
8. Have a serum creatinine greater than 2.0 mg/dl
9. Have hypersensitivity to ergocalciferol or any component of the formulation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2007-10 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Size of parathyroid glands | Baseline to 3-months post treatment
  Size of individual gland recorded while only the gland with maximum size at baseline included for analysis of primary endpoint. With sample size of 22, a two-sided 95% confidence interval for mean changes in size of parathyroid glands will extend 2.09 from observed mean, assuming that standard deviation is known to be 5 and confidence interval is based on the z statistic. Parameters for parathyroid glands compared pre- and post-replacement on an individual, gland-by-gland basis.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org